CLINICAL TRIAL: NCT02825719
Title: Pilot Study on the Pre-operative Use of Ulipristal on Fibroid in Chinese Population
Brief Title: Ulipristal Use in Chinese Population
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Ulipristal was withdrawal from the market
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Lui Man Wa, Dr, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 15-022
Record Dates: First submitted 2016-05-29; First posted 2016-07-07 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Fibroid
Keywords: Fibroid; Ulipristal; Selective progesterone receptor modulator; Chinese
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; ferrous sulfate; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ulipristal (Experimental): Patients will be prescribed Ulipristal acetate 5mg daily for 12 weeks before operation. If the patients have anaemia with haemoglobin less than 10g/dL, ferrous sulphate 300mg three times a day will be prescribed as well. Tranexamic Acid 500mg four times a day will be prescribed on request basis.
  Interventions: Drug: Ulipristal acetate; Drug: Ferrous sulphate; Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Patients will be prescribed placebo pills daily for 12 weeks before operation. If the patients have anaemia with haemoglobin less than 10g/dL, ferrous sulphate 300mg three times a day will be prescribed as well. Tranexamic Acid 500mg four times a day will be prescribed on request basis.
  Interventions: Other: Placebo pills; Drug: Ferrous sulphate; Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Ulipristal acetate — Ulipristal acetate 5mg daily will be prescribed
  Other Names: Esyma
  Arms: Ulipristal
Other: Placebo pills — Placebo pills will be prescribed
  Arms: Placebo
Drug: Ferrous sulphate — Ferrous sulphate 300mg three times a day will be prescribed if haemoglobin level is less than 10g/dL.
  Other Names: Ferasul
Drug: Tranexamic Acid — Tranexamic Acid 500mg four times a day on request basis will be prescribed if patient complained of menorrhagia.
  Other Names: Transamin

SUMMARY:
Uterine leiomyomas is the commonest benign tumour of the female genital tract. It lead to menorrhagia, anaemia, pain and pressure symptoms. Due to the enlarged uterus, the use of minimal invasive surgery is limited. There is also increase risk of intraoperative blood transfusion. Ulipristal acetate (UPA) is a selective progesterone-receptor modulator (SPRM). Preoperative use of Ulipristal for 12 weeks has been shown to decrease uterine bleeding, fibroid volume, pre-operative anaemia and symptoms severity. However there is still lacking evidence in terms of long term safety and efficacy, especially in Chinese population. The aim of the present study is to evaluate the effect and safety on preoperative use of Ulipristal on fibroid.

DETAILED DESCRIPTION:
Uterine leiomyomas is the commonest benign tumour of the female genital tract. It is often asymptomatic, but can also lead to anaemia, pain and pressure symptoms. It is the commonest indication for hysterectomy, especially abdominal hysterectomy. Currently, the use of hormonal treatment is associated with side effects including gastrointestinal upset, bloating, weight gain and thromboembolic risks. The main stay for treatment relies on surgery.

Furthermore, the use of minimal invasive surgeries is limited by the size of the fibroids. Preoperative use of Gonadotrophic Releasing Hormone analogues (GnRHa) is effective in shrinkage of the uterine leiomyomas and reduction of uterine bleeding. However, postmenopausal symptoms including hot flushes, vaginal dryness are profound.

Ulipristal acetate (UPA), previously named CDB-2914, is a selective progesterone-receptor modulator (SPRM). It binds to the progesterone receptors with high affinity. It inhibits follicular development and ovulation, while it has no significant effects on estradiol levels and antiglucocorticoid activity. Preoperative use of Ulipristal for symptomatic uterine fibroids has been investigated in randomized controlled study with improvement in terms of uterine bleeding, fibroids volume, pre-operative anaemia and symptoms severity. However there is still lacking evidence in terms of long term safety and efficacy. Also there is lack of evidence in Chinese population.

The aim of the present study is to evaluate the effect and safety on preoperative use of Ulipristal on fibroid.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for hysterectomy for symptomatic fibroid
* Be a Chinese
* Pre-menopausal
* With a Pictorial bleeding assessment chart score > 100 during menstruation at the preceding month
* Non-pregnant
* With a body-mass index between 18 to 30.

Exclusion Criteria:

* History of uterine surgery (apart from Caesarean section or cervical conization), endometrial ablation or uterine artery embolization
* History of gynaecological malignancies
* History of endometrial hyperplasia
* Known haemoglobinopathy (e.g. thalassaemia)
* Known severe coagulation disorder
* Has one or more ovarian cysts >= 4 cm in diameter diagnosed by ultrasound
* History of use of Selective Progesterone Receptor Modulator (SPRM)
* Current (within 12 months) problem with alcohol or drug abuse.
* Known allergy to SPRM or ferrous sulphate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change of uterine bleeding | Through study completion, an average of 14weeks
  Pictorial bleeding assessment chart will be used for assessment of uterine bleeding. Patients will be assessed before the start of treatment, after completion of 6 weeks course and after completion of 12 weeks course. The change of uterine bleeding after completion of 12 weeks course of treatment will be recorded.

SECONDARY OUTCOMES:
Change of haemoglobin level | Through study completion, an average of 14weeks
  The change of haemoglobin level after completion of 12 weeks course will be recorded.
Change of fibroid volume | Through study completion, an average of 14weeks
  The fibroid volume will be measured using ultrasonography before start of treatment, after 6 weeks course of treatment and after completion of 12 weeks course of treatment.
Intraoperative blood loss | After completion of 12 weeks course, the intraoperative blood loss at the time of performance of hysterectomy will be assessed.
  The amount of blood loss at hysterectomy will be recorded.
Conversion to less invasive intervention options | After completion of 12 weeks course of treatment and before the scheduled operation
  2 weeks before scheduled operation, patients will be assessed by the operation team and the most suitable route of hysterectomy will be discussed again. The possibility of conversion to less invasive intervention options including from laparotomy to laparoscopy will be recorded.
Side effects | Through study completion, an average of 14weeks
  The side effects including nausea, vomiting, headache, dyspepsia will be recorded.
Histology of the operative specimen | After completion of 12 weeks course of treatment
  Presence of malignancy or hyperplasia in the operative specimen will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest H. Y. Ng, Study Director — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
This is to protect the privacy of individual patients

REFERENCES:
- [Background] Parker WH. Etiology, symptomatology, and diagnosis of uterine myomas. Fertil Steril. 2007 Apr;87(4):725-36. doi: 10.1016/j.fertnstert.2007.01.093. PMID 17430732
- [Background] Jacobson GF, Shaber RE, Armstrong MA, Hung YY. Hysterectomy rates for benign indications. Obstet Gynecol. 2006 Jun;107(6):1278-83. doi: 10.1097/01.AOG.0000210640.86628.ff. PMID 16738152
- [Background] Jacoby VL, Autry A, Jacobson G, Domush R, Nakagawa S, Jacoby A. Nationwide use of laparoscopic hysterectomy compared with abdominal and vaginal approaches. Obstet Gynecol. 2009 Nov;114(5):1041-1048. doi: 10.1097/AOG.0b013e3181b9d222. PMID 20168105
- [Background] Lethaby A, Vollenhoven B, Sowter M. Pre-operative GnRH analogue therapy before hysterectomy or myomectomy for uterine fibroids. Cochrane Database Syst Rev. 2001;(2):CD000547. doi: 10.1002/14651858.CD000547. PMID 11405968
- [Background] Blithe DL, Nieman LK, Blye RP, Stratton P, Passaro M. Development of the selective progesterone receptor modulator CDB-2914 for clinical indications. Steroids. 2003 Nov;68(10-13):1013-7. doi: 10.1016/s0039-128x(03)00118-1. PMID 14667994
- [Background] Nieman LK, Blocker W, Nansel T, Mahoney S, Reynolds J, Blithe D, Wesley R, Armstrong A. Efficacy and tolerability of CDB-2914 treatment for symptomatic uterine fibroids: a randomized, double-blind, placebo-controlled, phase IIb study. Fertil Steril. 2011 Feb;95(2):767-72.e1-2. doi: 10.1016/j.fertnstert.2010.09.059. Epub 2010 Nov 5. PMID 21055739
- [Result] Donnez J, Tatarchuk TF, Bouchard P, Puscasiu L, Zakharenko NF, Ivanova T, Ugocsai G, Mara M, Jilla MP, Bestel E, Terrill P, Osterloh I, Loumaye E; PEARL I Study Group. Ulipristal acetate versus placebo for fibroid treatment before surgery. N Engl J Med. 2012 Feb 2;366(5):409-20. doi: 10.1056/NEJMoa1103182. PMID 22296075